CLINICAL TRIAL: NCT04148768
Title: Acute Effect of Inferential Therapy (IFT) and Short Wave Diathermy (SWD) on Balance in Subjects With Knee Pain
Acronym: IFT & SWD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Snehil Dixit, Assistant Professor , Department of Medical Rehabilitation, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (ECM#2019-55)-( HAPO-06-B-001)
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Knee Acute and Chronic Pain
Keywords: Knee pain; osteoarthritis,; patello-femoral pain,; Anetrior cruciate repair; Balance; Dynamic and static balance; Proprioception
MeSH Terms: conditions — Chronic Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Intervention SWD & IFT: 4 SESSIONS OF TREATMENT and measurement of balance
Who Masked: Participant
Masking Description: Participants will not be aware of the treatment groups given to them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferential therapy (Active Comparator): Interferential therapy will be given using 4 electrode methods. The 'medium frequency' currents (medium frequency in electromedical terms is usually considered to be 1KHz-100KHz). These medium frequency currents, passed through the tissues simultaneously, where they are set up so that their paths cross & they literally interfere with each other. This interaction gives rise to an interference current (or beat frequency) which has the characteristics of low-frequency stimulation. Pre-Post Y balance test will be used after 4 sessions to measure the improvement in balance in the population
  Interventions: Device: Inferential therapy
- Shortwave diathermy (Active Comparator): 4 sessions of treatment will be given to the participants with SWD. Pre-post Y balance test will be used to measure balance in the population
  Interventions: Device: short wave diathermy

INTERVENTIONS:
Device: Inferential therapy — Interferential therapy(IFT) utilises two of these medium frequency currents, passed through the tissues simultaneously, where they are set up so that their paths cross & they literally interfere with each other - hence another term that has been used in the past but appears to be out of favour at the moment - Interference Current Therapy. This interaction gives rise to an interference current (or beat frequency) which has the characteristics of low-frequency stimulation.
  Arms: Inferential therapy
Device: short wave diathermy — SWD: Technical specification of Generator frequency: 27.12 MHz, ± 0.6% Output power: continuous High-Frequency max. 400 W, pulsed High-Frequency max. 1000 W (peak) Pulse duration: ca. 400 µs Pulse repetition frequency: 15-200 Hz adjustable in 10 steps Mains supply: 230-240 V / 50 Hz Mains voltage variation: approx. ± 10% Current consumption: approx. 6 Ampere (at 230 V)
  Arms: Shortwave diathermy

SUMMARY:
Background: The Y balance test is a dynamic test that requires strength, flexibility, and proprioception. It is a measure of dynamic balance that provides a significant challenge to athletes and physically active individuals. The test can be used to assess physical performance, but can also be used to screen deficits in dynamic postural control due to musculoskeletal injuries (e.g. chronic ankle instability), to identify athletes at greater risk for lower extremity injury, as well as during the rehabilitation of orthopedic injuries in healthy active adults

Objective: To know the effect of 4 sessions of treatment by interferential therapy (IFT) 15-20 minutes, and SWD 15 min on the balance and dynamic postural component using Y balance test

Methods: Subjects will be randomized into IFT and laser group (n=20 each). After the first session, the balance component will be measured pre-post-intervention.

Outcome assessment: Y Balance tests score.

DETAILED DESCRIPTION:
Objective: To know the effect of 4 sessions of treatment by interferential therapy, and SWD on the balance and dynamic postural component using Y balance test

Methods:

Study design: Random sampling through lottery methods Blinding: Participants were not aware of the group they were in Allocation concealment: Not done Inclusion criteria: Physical assessment of the knee joint participants complains of pain, osteoarthritis, Patellofemoral knee pain syndrome, pain due to altered biomechanics of knee joints (structural and functional) Exclusion criteria: History of previous surgeries, participants on steroids, Vitamin deficiencies, osteoporosis, open wounds, recurrent ACL repair, Affliction due to metastasis or post-cancer patients

Treatment specifications:

Duration of intervention: Treatment will continue for 4 sessions/week, with each session lasting 15-20 minutes.

Intervention:

Experimental group-1: Interferential therapy will be given to the patients with knee pain for 4 sessions for 15-20 minutes and the examination of the balance will be done with Y balance tests Pre-Post. 4 electrodes methods placed diagonally to each other creating a beat frequency at the center. Intensity to the percieved tolerable limits. The 'medium frequency' currents (medium frequency in electromedical terms is usually considered to be 1KHz-100KHz). These medium frequency currents, passed through the tissues simultaneously, where they are set up so that their paths cross & they literally interfere with each other. This interaction gives rise to an interference current (or beat frequency) which has the characteristics of low-frequency stimulation

Experimental group-2: SWD will be given to the patients with knee pain for 4 sessions for 10-15 minutes with Continuous Mode and intensity: comfortable warmth, timing 15 mins and examination of the balance will be done with Y balance tests Pre-Post.

Technical specification : Technical specification of Generator frequency: 27.12 MHz, ± 0.6% Output power: continuous High-Frequency max. 400 W, pulsed High-Frequency max. 1000 W (peak) Pulse duration: ca. 400 µs Pulse repetition frequency: 15-200 Hz adjustable in 10 steps Mains supply: 230-240 V / 50 Hz Mains voltage variation: approx. ± 10% Current consumption: approx. 6 Ampere (at 230 V) Dimensions (width, without arms): 56x43x92.5 cm Length electrode arms: 93 cm Weight: ca. 80 kg.

ELIGIBILITY:
Inclusion Criteria:

1. Non-specific Knee pain,
2. osteoarthritis,
3. chronic ACL and meniscus injury,
4. patellofemoral knee pain

Exclusion Criteria:

1. Recent major surgeries within 6 months,
2. Limb Length discrepancies, amputation,
3. any musculoskeletal or neurological limitation preventing evaluation,
4. vitamin deficiency (B12),
5. neuropathy,
6. cancer-related patients,
7. rheumatoid arthritis,
8. Osteoporosis

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-04-27 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Y balance test Score | Change is being evaluated from Baseline and at 4 week
  More condensed form of star excursion test. Used to evaluate dynamic balance

SECONDARY OUTCOMES:
Visual analogue scale | Change is being evaluated from Baseline and at 4 week
  Pain values from 0-10 on a scale 0 means no pain 10 means maximum unbearable pain

CONTACTS AND LOCATIONS:
Overall Officials: snehil dixit, PhD, Principal Investigator — King Khalid University
Locations (1):
- King Khalid University, Abhā, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided